CLINICAL TRIAL: NCT02831816
Title: Clinical Evaluation of ZP, A Patient Preoperative Skin Preparation
Brief Title: Clinical Evaluation of Patient Preoperative Prep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZX-ZP-0074 / 150316-103
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Surgical Skin Preparation
MeSH Terms: interventions — citrate, isopropyl alcohol, methylene blue, parabens drug combination; Ethanol; Chromogranins; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZP (70% IPA) (Experimental): Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ZuraPrep
- ChloraPrep (Active Comparator): Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  Interventions: Drug: ChloraPrep
- ZP Vehicle (Placebo Comparator): ZP without IPA
  Interventions: Drug: ZP Vehicle

INTERVENTIONS:
Drug: ZuraPrep — Apply topically.
  Other Names: Isopropyl alcohol 70%; ZP
  Arms: ZP (70% IPA)
Drug: ChloraPrep — Apply topically.
  Other Names: CHG 2% / IPA 70%; Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Arms: ChloraPrep
Drug: ZP Vehicle — Apply topically.
  Other Names: ZP without IPA
  Arms: ZP Vehicle

SUMMARY:
The objective of the study is to demonstrate the antimicrobial efficacy of the ZP Preoperative Prep on skin flora of the abdomen and inguinal regions of human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race.
* Subjects in good health.
* Minimum skin flora baseline requirements on abdomen and groin.
* Skin free of tattoos, dermatoses, abrasions, cuts, lesions, or other skin disorder near or on the applicable test area.

Exclusion Criteria:

* Topical or systemic antimicrobial exposure within 14 days prior to screening and treatment days, including antibiotics.
* Subjects with a history of skin sensitivity, skin allergies, or skin cancer.
* Subjects who are pregnant, attempting pregnancy, or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BioScience Laboratories, Inc., Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edmiston CE, Lavin P, Spencer M, Borlaug G, Seabrook GR, Leaper D. Antiseptic efficacy of an innovative perioperative surgical skin preparation: A confirmatory FDA phase 3 analysis. Infect Control Hosp Epidemiol. 2020 Jun;41(6):653-659. doi: 10.1017/ice.2020.27. PMID 32131912

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment consists of subjects that advanced from screening to randomization and treatment. Each subject had 2 test products applied bilaterally; therefore, the numbers will not add up uniformly across arms due to the pre-determined cohort/block design. Result totals will be less than than the treated number as the per subject/ area/intervention anatomical site must have an acceptable baseline count/flora.
Units Other Than Participants: Ab or groin
Groups:
- All Participants: ZP (Isopropyl alcohol (IPA) 70%) or CP or ZP Vehicle
  Applied topically to ab (for 30 seconds) or groin (for 2 minutes).
Period: Overall Study
Arm/Group | All Participants
Started | 640; 640 Ab or groin
ZP | 589; 589 Ab or groin
CP | 590; 590 Ab or groin
Vehicle | 131; 131 Ab or groin
Completed | 640; 640 Ab or groin
Not Completed | 0; 0 Ab or groin

BASELINE CHARACTERISTICS:
Groups:
- Treated Population: Each subject could have received 2 out of 3 test products randomly assigned. Demographics were not stratified by test product due to study design. While 640 was the treated population, to be evaluable for efficacy, each subject anatomical sample site (4/per subject) would need to pass the minimum log10 cfu/cm^2 baseline requirements.
Arm/Group | Treated Population
Number analyzed (Participants) | 640
Age, Continuous [Median (Full Range); unit: years] | 30 [18 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 476
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 581
  Unknown or Not Reported | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 576
  More than one race | 0
  Unknown or Not Reported | 32

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Reduction
Description: A a 3-log per cm2 bacterial reduction on the inguinal region is considered a success.
Time Frame: 10 minutes post product application
Population: Treated subjects with treatment day baseline criteria 5.0-7.5 log recoveries.
Measure: Mean (Standard Deviation); unit: log10 cfu/cm^2
Groups:
- Mean Log Reduction - ZP (70% IPA) - Groin: Isopropyl alcohol (IPA) 70%
  ZuraPrep: Apply topically to groin.
- Mean Log Reduction - Groin - ChloraPrep: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically to groin.
- Mean Log Reduction - Groin - ZP Vehicle: ZP without IPA
  ZP Vehicle: Apply topically to the groin.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Groin | Mean Log Reduction - Groin - ChloraPrep | Mean Log Reduction - Groin - ZP Vehicle
Number analyzed (Participants) | 342 | 352 | 74
log10 cfu/cm^2 | 4.04 (1.33) | 4.01 (1.43) | 1.60 (0.69)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - Groin - ChloraPrep; Groin 10 minutes Average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 cfu/cm2 less than the active control; Median Difference (Final Values) = -0.020, 95% CI 2-sided [-0.221 to 0.180]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Groin vs Mean Log Reduction - Groin - ZP Vehicle; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Median Difference (Final Values) = 2.45, 95% CI 2-sided [2.15 to 2.76]

2. Primary Outcome: Bacterial Reduction - Abdomen
Description: A 2-log per cm2 bacterial reduction on the abdomen region is considered a success.
Time Frame: 10 minutes post product application
Population: Treated subjects with treatment day baseline criteria 3.0-5.5 log10 recoveries.
Measure: Mean (Standard Deviation); unit: log10 cfu/cm^2
Groups:
- Mean Log Reduction - ZP (70% IPA) - Abdomen: Isopropyl alcohol (IPA) 70%
  ZuraPrep: Apply topically to abdomen.
- Mean Log Reduction - Abdomen - ChloraPrep: Chlorhexidine gluconate (CHG) 2% / Isopropyl alcohol (IPA) 70%
  ChloraPrep: Apply topically to Abdomen.
- Mean Log Reduction - Abdomen - ZP Vehicle: ZP without IPA
  ZP Vehicle: Apply topically to the Abdomen.
Arm/Group | Mean Log Reduction - ZP (70% IPA) - Abdomen | Mean Log Reduction - Abdomen - ChloraPrep | Mean Log Reduction - Abdomen - ZP Vehicle
Number analyzed (Participants) | 324 | 320 | 68
log10 cfu/cm^2 | 2.99 (1.1) | 2.79 (1.1) | 1.00 (0.9)
Statistical Analysis 1: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - Abdomen - ChloraPrep; Abdomen 10 minutes average treatment effect, calculated using a linear regression model for each body site, was used for primary analysis. In the model, the response was the post-treatment log10 bacterial counts and predictors were the treatment effect as a fixed effect and the pre-treatment log10 bacterial counts as a covariate; Test type: Non-Inferiority — Investigational product cannot be more than 0.05 log10 cfu/cm2 less than the active control; Mean Difference (Final Values) = -0.0435, 95% CI 2-sided [-0.2085 to 0.1215]
Statistical Analysis 2: Comparison: Mean Log Reduction - ZP (70% IPA) - Abdomen vs Mean Log Reduction - Abdomen - ZP Vehicle; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [1.70 to 2.25]

ADVERSE EVENTS:
Time Frame: 6 hours post product application
Arm/Group | ZP (70% IPA) | ChloraPrep | ZP Vehicle
All-Cause Mortality (participants affected / at risk) | 0/589 | 0/590 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/589 | 0/590 | 0/131
Other Adverse Events (participants affected / at risk) | 0/589 | 0/590 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02831816/Prot_SAP_000.pdf